CLINICAL TRIAL: NCT06229977
Title: A Randomized Controlled Trial of the Fatty Acid Amide Hydrolase Inhibitor Palmitoylethanolamide in Bipolar Depression
Brief Title: A Trial of the Fatty Acid Amide Hydrolase Inhibitor Palmitoylethanolamide in Bipolar Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Baszucki Brain Research Fund (Other)
Responsible Party: Principal Investigator, Rodrigo Machado-Vieira, MD, PhD, MSc, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC-MS-21-0989
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Bipolar Depression
Keywords: cytokine levels
MeSH Terms: conditions — Bipolar Disorder | interventions — palmidrol; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PEA plus Treatment as Usual (TAU) (Experimental)
  Interventions: Drug: Palmitoylethanolamide (PEA); Drug: Treatment as Usual (TAU)
- Placebo plus Treatment as Usual (TAU) (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Treatment as Usual (TAU)

INTERVENTIONS:
Drug: Palmitoylethanolamide (PEA) — Participants will receive PEA at a dose of 600mg twice daily for 6 weeks.
  Arms: PEA plus Treatment as Usual (TAU)
Drug: Placebo — Participants will receive placebo (a tablet that contains no active ingredient) to be taken twice daily for 6 weeks
  Arms: Placebo plus Treatment as Usual (TAU)
Drug: Treatment as Usual (TAU) — subjects will receive a mood stabilizer per usual care

SUMMARY:
The purpose of this study is to o evaluate the antidepressant efficacy of the PEA in Bipolar Depression and the association between antidepressant response with endogenous cannabinoids and cytokine levels

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Bipolar Disorder according to the Diagnostic and Statistical Manual of Mental Disorders (Structured Clinical Interview), Fifth Edition, (DSM5), with a score of ≥16 on the 17-item HAM-D
* currently in use of at least one FDA approved mood stabilizer with or without antidepressant
* medically and neurologically healthy on the basis of medical history, physical examination

Exclusion Criteria:

* Cannabis misuse according to clinical judgement
* unstable medical condition or uncontrolled medical problem with known central nervous system (CNS) effects
* active DSM-5 substance use disorder in past three months (other than alcohol or nicotine use disorder)
* acute high suicidal risk
* in a manic episode
* current psychotic features or cognitive impairment that would preclude understanding of the consenting process or tests/examination
* pregnant or nursing women
* unstable medical conditions
* clinically significant abnormal laboratory tests based on complete blood count, liver and kidney function when available

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-05-17 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2025-07-17 (Actual)

PRIMARY OUTCOMES:
Change in depression as assessed by the Hamilton Depression rating Scale (HAM-D) | Baseline, 6 weeks follow up
  This is a 13 item questionnaire and each is scored from 0-2 for a maximum score of 26 , a higher score indicating worse outcome

SECONDARY OUTCOMES:
Percentage of participants that show a remission of depressive symptoms as assessed by the HAM-D scale. | from baseline to end of study (6 week follow up)
  Remission of depressive symptoms are defined by a score of ≤7 on the HAM-D. This is a 13 item questionnaire and each is scored from 0-2 for a maximum score of 26 , a higher score indicating worse outcome
Percentage of participants that show a response as assessed by the HAM-D scale | from baseline to end of study (6 week follow up)
  Response rate is defined by ≥ 50 % reduction in depression score(HAM-D). This is a 13 item questionnaire and each is scored from 0-2 for a maximum score of 26 , a higher score indicating worse outcome
Number of participants that show early improvement as defined by >20% improvement in HAM-D depression score | From baseline to week 2 visit
  This is a 13 item questionnaire and each is scored from 0-2 for a maximum score of 26 , a higher score indicating worse outcome
Change in depression as assessed by the Montgomery Äsberg Depression Rating Scale (MADRS) | Baseline, 6 weeks follow up
  This is a 10 item questionnaire and each is scored from 0 -6 for a maximum score of 60, higher score indicating worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Machado-Vieira, M.D, Ph.D., M.Sc, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No